CLINICAL TRIAL: NCT02055469
Title: Achalasia; Mechanisms Underlying Persistent Symptoms After Treatment
Brief Title: Achalasia: Mechanisms Underlying Treatment Failure
Status: Terminated | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 009393
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Achalasia
Keywords: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In patients with achalasia, the relationship between the perception of dysphagia, oesophageal emptying, lower oesophageal sphincter (LOS) distensibility and oesophageal circular and longitudinal muscle contraction is not clear.

We aim to characterize oesophageal circumferential and longitudinal muscle contractility and LOS distensibility in patients with achalasia (either before or after treatment). This may allow an understanding of the mechanisms underlying persistent dysphagia and delayed oesophageal emptying after treatment.

DETAILED DESCRIPTION:
This is observational study of patients with achalasia (with or without treatment). Treatment will have been a previous Heller's myotomy or pneumatic dilatation (and is not randomised). Patients with known or suspected achalasia will attend the GI physiology unit at the Royal London Hospital for standard care. Standard care involves assessing the perception of dysphagia with questionnaires, assessing oesophageal circular muscle function with high resolution oesophageal manometry (HRM) and oesophageal emptying with a timed barium oesophagram (TBO). The two experimental tests performed as part of the study (which are not currently routine care) are EndoFLIP and HFIUS.

On arrival at the GI physiology unit, patients will be given verbal and written information about the study (including standard care and non-standard tests). They will then be asked if they wish to participate. Informed written consent will be obtained.

Participants will complete questionnaires and HRM. If HRM is not consistent with achalasia, the patient's participation in the study ends. If HRM is consistent with achalasia then the participant will then undergo EndoFLIP, HFIUS and TBO.

Assessments are as follows (but are not necessarily done in the order given:

A. Perception of dysphagia (using MAYO and Eckardt questionnaires)

Dysphagia questionnaires are a non-intrusive, quick and well validated method of assessing the perception of dysphagia and are considered part of standard care.

B. Oesophageal circular muscle function (using HRM)

HRM is part of standard care and is performed in the GI physiology unit routinely by appropriately trained and experienced investigators. It involves the insertion of a small catheter into the oesophagus via the transnasal route. The only risk to the patient is nasopharyngeal discomfort on insertion, which is reduced by the use of nasal lignocaine spray. Ten 5ml water swallows are assessed and the duration is typically 10 to 15 minutes.

C. Oesophageal emptying (using TBO)

TBO is a standard/routine investigation in assessing suspected or treated achalasia. It is a variant of a "barium swallow". The patient drinks 200mls of barium and has plain radiological films taken at 1,3 and 5 minutes. The TBO is performed in the GI physiology unit by investigators with appropriate training and certification (IRMER). It involves the use of ionising radiation (X rays) but is not an experimental procedure.

D. Distensibility of the mid oesophagus and LOS (using EndoFLIP)

Endoscopic functional luminal imaging probe (EndoFLIP) is not part of standard care. It is very similar to HRM as it uses a small catheter which is inserted into the oesophagus via the transnasal route. There is a small water filled balloon at the tip of the catheter which is gently inflated using water. The distensibility of any part of the oesophagus is thus able to be measured. Like HRM the only risk to the participant is nasopharyngeal discomfort on insertion. The duration of the procedure is 10 to 15 minutes.

E. Longitudinal muscle thickness and contraction (using HFIUS)

High frequency intra luminal ultrasound (HFIUS) is not part of standard care and will be performed in the endoscopy unit of the Royal London Hospital (which is located very close to the GI physiology unit). Like HRM and EndoFLIP, it uses a small catheter which is inserted into the oesophagus via the transnasal route. It is able to visualise the layers of the oesophageal wall. Again, the only risk to the patient is discomfort. The procedure takes about 10 to 15 minutes.

Patients with achalasia will classified on TBO as having either normal or delayed oesophageal emptying. The perception of dysphagia and motility characteristics of these two groups will then be compared using an independent samples t test. SPSS will be used for statistical analysis. An independent statistician has reviewed and approved the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with achalasia diagnosed on HRM criteria, with or without previous treatment
* Written ICF signed voluntarily before the first trial-related activity.
* Male or female, aged 18-70
* If the subject is a woman of childbearing potential, she must have a negative urine pregnancy test before the start of assessments

Exclusion Criteria:

* Any abnormal oesophageal motility finding that is not consistent with achalasia
* History of gastrointestinal tract surgery, fundoplication, endoscopic anti reflux procedure or any other recent abdominal operation in the last 6 months
* Major psychiatric, neurological, respiratory, liver, haemorrhagic and cardiac disorders, malignancies
* Pregnancy
* Subjects with a documented history of long segment (>3 cm) Barrett's oesophagus, large (> 3 cm) hiatus hernia, structural abnormalities of oesophagus (i.e. Rings, webs, scleroderma)
* Use of prokinetic medication less than 7 days before the start of the study
* Any condition that in the opinion of the Investigator would complicate or compromise the trial or the well-being of the subject.
* Evidence of any clinically relevant pathology that could interfere with trial results or put subject safety at risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with achalasia (or suspected achalasia) either before or after treatment referred from secondary care to the GI physiology unit of the Royal London Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Perception of dysphagia | Baseline (At recruitment )
  Questionnaires
Oesophageal circumferential muscle contractility | Baseline (At recruitment )
  Using high resolution oesophageal manometry
Oesophageal longitudinal muscle contraction | Baseline (At recruitment )
  High frequency intraluminal oesophageal ultrasound
Oesophageal emptying | Baseline (At recruitment )
  Timed barium oesophagram
Assessment of oesophageal and LOS distensibility | Baseline (At recruitment )
  Using endoscopic functional luminal imaging probe (EndoFLIP)

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, UK, United Kingdom